CLINICAL TRIAL: NCT04094883
Title: Institute for Global Health and Infectious Diseases (IGHID) 11911 - Cross-reactive N. Gonorrhoeae Immune Responses Induced by a N. Meningitidis Vaccine
Brief Title: Study to Assess Gonorrhoeae Immune Responses Induced by a N. Meningitidis Vaccine
Acronym: 4CMenB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-1145
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Results first posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Neisseria Gonorrhoeae Infection
Keywords: Neisseria gonorrhoeae; Cross-reactive; Immune; Responses; Neisseria meningitidis; Vaccine
MeSH Terms: conditions — Gonorrhea | interventions — 4CMenB vaccine

STUDY DESIGN:
Intervention Model Description: All participants will receive the group B meningitis vaccine (brand name Bexsero™).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 4CMenB Vaccine (Experimental): Participants will receive the 4CMenB (Bexsero) vaccine by an injection in the deltoid region of the upper arm or the higher front area on one side of the thigh at the enrollment visit (Day 0) and at week 5.
  Interventions: Biological: Meningococcal Group B Vaccine

INTERVENTIONS:
Biological: Meningococcal Group B Vaccine — All participants will receive the 4CMenB vaccine, 0.5 mL, at entry (Day 0) and at week 5.
  Other Names: Bexsero; 4-component Neisseria meningitidis group B vaccine; 4CMenB

SUMMARY:
The purpose of this study is to test whether the group B meningitis vaccine (brand name Bexsero™) induces immune responses against the bacteria that causes gonorrhea.

Participants: Approximately 15 Individuals who are 18-25 years of age that are not pregnant, HIV negative, have no history of congenital immunologic disorder, and are not taking immune suppressive medications will be enrolled on this study at a single site, University of North Carolina at Chapel Hill (UNC-CH).

Procedures (methods): Participants will receive two-doses of an FDA-approved vaccine that provides protection from N. meningitidis infection according to the recommended dosing schedule. The first vaccine dose will be given to participants at the entry visit and the second vaccine dose will be given to participants at the week 5 visit. The participants will provide samples of blood as well as mucosal surface derived samples (urine and/or swabs) at four separate visits (entry, week 5, week 6, and week 7).

DETAILED DESCRIPTION:
This study is a single center, single arm, interventional pilot study in which participants will receive two-doses of the 4CMenB vaccine according to the recommended administration schedule and will provide blood, pharyngeal swabs, and urine or self-collected vaginal swabs at each of four study visits.

The study population will include 15 individuals aged 18-25 years with no contraindication to vaccination and no known immune compromising medical condition or medication.

Participants will be seen for informed consent and eligibility screening. Enrolled participants will be given 1 dose of 4CMenB at enrollment and a second dose at week 5. Participants will be seen at entry, weeks 5, 6, and 7 for blood collection, pharyngeal swabs, and provide urine (male participants) or self-collected vaginal swabs collected for secondary screening and baseline immunologic testing.

Screening Evaluations Screening evaluations include: medical history, medication history within the past 60 days, vital signs, targeted physical exam, and pregnancy test for female participants of child bearing potential). Screening visit must be conducted no greater than 30 days prior to enrollment visit. The screening evaluation and enrollment visit can all occur on the same day. Participants may be re-screened one time.

Entry Evaluations

Entry evaluations will be collected PRIOR to phlebotomy, specimen collection, and vaccine administration:

Acute Illness Assessment will be completed before phlebotomy, specimen collection, and vaccine administration. Participants who have an acute illness may be rescheduled for their phlebotomy, specimen collection, and vaccine within their screening visit window.

Update medical history and concomitant medications. Conduct a targeted physical exam and collect vital signs [heart rate (HR), blood pressure (BP), oral temperature (Temp), respiration rate (RR), and weight] prior to phlebotomy to collect up to 60 mL of blood, specimen collection, and vaccine administration.

For females of reproductive potential, negative urine pregnancy testing results must be available before phlebotomy, specimen collection, and vaccine administration.

Samples to be stored for immunologic testing will be batch run at the end of the study:

pharyngeal swabs, urine sample (from male participants), self-collected vaginal swabs (from female participants), serum, and peripheral blood mononuclear cells (PBMC).

Post-Entry Evaluations

Week 5 Evaluations:

Acute Illness Assessment will be completed before phlebotomy, specimen collection, and vaccine administration. Participants who have an acute illness or who have taken exclusionary anticoagulant medications may be rescheduled for their vaccine within their screening visit window.

Update medical history and concomitant medications before phlebotomy and vaccine administration. Conduct a targeted physical exam and collect vital signs (HR, BP, Temp, RR) before phlebotomy to collect up to 60 mL of blood, specimen collection, and vaccine administration.

For females of reproductive potential, negative urine pregnancy testing results must be available before phlebotomy, specimen collection, and vaccine administration.

Week 5 laboratory evaluations will be collected PRIOR to vaccine administration:

Samples to be stored for immunologic testing will be batch run at the end of the study:

pharyngeal swabs, urine sample (from male participants), self-collected vaginal swabs (from female participants), serum, and PBMC.

Week 6 and Week 7 Evaluations:

Update medical history and concomitant medications prior to phlebotomy to collect up to 60 mL of blood and specimen collection.

Samples to be stored for immunologic testing will be batch run at the end of the study:

pharyngeal swabs, urine sample (from male participants), self-collected vaginal swabs (from female participants), serum, and PBMC.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and give informed consent
2. Willingness to undergo all study procedures.
3. Males or females between the ages of 18 to 25 at screening (inclusive).
4. Good health, as determined by medical history and targeted physical exam.
5. Participants agree to abstain from vaccines from study entry to 30 days after receipt of the second 4CMenB vaccine.
6. Female participants of child bearing potential must have a negative urine pregnancy test at the screening visit, and prior to receipt of vaccines at study entry and week 5 visits. Self-reported history is acceptable documentation of hysterectomy, bilateral oophorectomy, tubal ligation, or tubal micro-inserts which eliminate child bearing potential of participant. If participating in sexual activity that could lead to pregnancy, women must agree to use a form of contraceptive until 28 days after completion of the vaccine series. At least one of the following methods must be used appropriately: Condoms (male) with or without spermicidal agent, Diaphragm or cervical cap with spermicide, Intrauterine device (IUD), or Hormone-based contraceptive. Self-report of a monogamous male partner who has a vasectomy is also acceptable.

Exclusion Criteria:

1. Known allergy/sensitivity or any hypersensitivity to latex or any of the components of the study product or its formulation (see section 5.2 for a list of components).
2. Participants who have received any vaccine directed against N. meningitidis serogroup B
3. Serious illness or injury requiring hospitalization within 21 days prior to study entry.
4. Current or prior history of a medical condition resulting in impaired immunity (such as HIV infection, inborn or acquired immunodeficiency syndromes, all cancers including leukemia or lymphoma, or the of use antineoplastic drugs or radiation treatment).
5. Known active infection with HIV, Hepatitis C Virus (HCV ), or Hepatitis B Virus (HBV). This information will be obtained verbally from the participant.
6. History of excessive alcohol consumption, drug abuse, psychiatric conditions, social conditions or occupational conditions that in the opinion of the investigator would preclude compliance with the study.
7. Hemophilia or other bleeding diatheses.
8. Receipt of anticoagulants (aspirin or nonsteroidal anti-inflammatory drugs (NSAIDS) are acceptable) within 14 days prior to study entry.
9. Autoimmune disorders; mild autoimmune disorders, such as eczema, are not exclusionary and will be determined by the investigator.
10. Use of any systemic immunomodulatory treatment, systemic corticosteroids, (inhaled and topical corticosteroids acceptable), investigational products, interleukins, interferons, growth factors, or intravenous immunoglobulin (IVIG) within 45 days prior to study entry.
11. Pregnant women and nursing mothers or women who are planning to become pregnant or breastfeed within 28 days after receipt of their second 4CMenB vaccine.
12. Have received any licensed vaccine within 30 days prior to study vaccination.
13. Have donated blood or blood products within 30 days before study vaccination, plan to donate blood at any time during the study and up to 30 days after the last blood draw.
14. Any condition in the opinion of the investigator that would interfere with the proper conduct of the trial.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Duncan, MD, PhD, Principal Investigator — UNC-Chapel Hill
Locations (1):
- University of North Carolina Health Care, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data that supports the results will be shared beginning 12 to 24 months following publication provided the investigator/researcher who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12-24 months after publication
Access Criteria: Other investigators/researchers who propose to use the individual participant data (IPD) from this study will need to have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and execute a data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 4CMenB Vaccine
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | 4CMenB Vaccine
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Anti-N. Gonorrhoeae Outer-membrane Vesicle Specific Immunoglobulin G (IgG) Concentrations After Immunization
Description: The change in concentrations presented as the difference in geometric mean concentration in human serum of IgG binding to N. gonorrhoeae strain FA1090 surface antigens Outer-membrane vesicles (OMV) determined by ELISA in serum from entry visit and week 7 visit
Time Frame: pre-vaccination at entry visit (prior to first vaccination, Day 0) and week 7 visit (2 weeks after second vaccination)
Measure: Geometric Mean (80% Confidence Interval); unit: titers
Arm/Group | 4CMenB Vaccine
Number analyzed (Participants) | 10
titers
  Anti-N. gonorrhoeae OMV titer (dilution giving half maximal response) - Entry Visit | 61.57 [38.7 to 97.97]
  Anti-N. gonorrhoeae OMV titer (dilution giving half maximal response) - Week 7 Visit | 206.2 [141.9 to 299.5]

2. Primary Outcome: Change in Anti-N. Gonorrhoeae Outer-membrane Vesicle Specific Immunoglobulin M (IgM) Concentrations After Immunization
Description: The change in concentrations presented as the difference in geometric mean concentration in human serum of IgM binding to N. gonorrhoeae strain FA1090 surface antigens (Outer-membrane vesicles) determined by ELISA in serum from entry visit and week 7 visit
Time Frame: pre-vaccination at entry visit (prior to first vaccination, Day 0) and week 7 visit (2 weeks after second vaccination)
Measure: Geometric Mean (80% Confidence Interval); unit: titer
Arm/Group | 4CMenB Vaccine
Number analyzed (Participants) | 10
titer
  Anti-N. gonorrhoeae OMV titer (dilution giving half maximal response) - Entry Visit | 86.89 [58.96 to 128.1]
  Anti-N. gonorrhoeae OMV titer (dilution giving half maximal response) - Week 7 Visit | 83.84 [57.34 to 122.6]

3. Primary Outcome: Change in Anti-N. Gonorrhoeae Outer-membrane Vesicle Specific Immunoglobulin A (IgA ) Concentrations After Immunization
Description: The change in concentrations presented as the difference in geometric mean concentration in human serum of IgA binding to N. gonorrhoeae strain FA1090 surface antigens (Outer-membrane vesicles) determined by ELISA in serum from entry visit and week 7 visit
Time Frame: pre-vaccination at entry visit (prior to first vaccination, Day 0) and week 7 visit (2 weeks after second vaccination)
Measure: Geometric Mean (80% Confidence Interval); unit: titer
Arm/Group | 4CMenB Vaccine
Number analyzed (Participants) | 10
titer
  Anti-N. gonorrhoeae OMV titer (dilution giving half maximal response) - Entry Visit | 3.689 [2.155 to 6.315]
  Anti-N. gonorrhoeae OMV titer (dilution giving half maximal response) - Week 7 Visit | 4.725 [3.044 to 7.335]

4. Primary Outcome: Mean Change in Proportion of Cluster of Differentiation 4 Positive (CD4+) T Cells Expressing at Least Two Different Activation Markers After Immunization
Description: Flow cytometry used to measure the number of CD4+ lymphocytes expressing Interferon-gamma (IFN-g), Tumor Necrosis Factor-alpha (TNF-a), Interleukin-2 (IL-2), and Cluster of Differentiation 107a (CD107a) after in vitro stimulation with N. gonorrhoeae strain FA1090 Outer-membrane vesicles in circulating peripheral blood mononuclear cells (PBMC). The frequency of CD4+ T cells expressing at least two activation markers will be expressed as a proportion of total CD4+ lymphocytes. The change in frequency will be presented as the difference between frequency of cells measured at entry visit and at week 7 visit.
Time Frame: pre-vaccination at entry visit (prior to first vaccination, Day 0) and week 7 visit (2 weeks after second vaccination)
Measure: Mean (80% Confidence Interval); unit: proportion CD4 cells
Arm/Group | 4CMenB Vaccine
Number analyzed (Participants) | 10
proportion CD4 cells
  proportion of CD4+ positive lymphocytes expressing least two activation markers -Entry Visit | 0.002750 [0.001222 to 0.004279]
  proportion of CD4+ positive lymphocytes expressing least two activation markers - week 7 Visit | 0.003058 [0.002552 to 0.003564]

ADVERSE EVENTS:
Time Frame: From signing of Informed Consent until study completion, a total of up to 26 weeks.
Arm/Group | 4CMenB Vaccine
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4CMenB Vaccine (N=11)
injection site (left deltoid) pain (General disorders) | 8 (16)
Injection site (left deltoid) tenderness (General disorders) | 4 (7)
Injection site (left deltoid) erythema (General disorders) | 2 (2)
Injection site (left deltoid) induration (General disorders) | 2 (2)
Injection site (left deltoid) swelling (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (4)
Subjective fever (General disorders) | 2 (2)
chills (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (5)
lightheadedness (Nervous system disorders) | 1 (1)
flushing (General disorders) | 1 (1)
pharyngitis (Infections and infestations) | 1 (1)
cough and nasal congestion (Infections and infestations) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 1 (1)
wisdom teeth extraction (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/83/NCT04094883/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/83/NCT04094883/ICF_001.pdf